CLINICAL TRIAL: NCT05475431
Title: The Most Appropriate Prescription of the First-line, the Second-line, and the Third Treatment for H. Pylori Eradication Among Patients Who Are Comorbid Diabetes Mellitus, Chronic Obstructive Pulmonary Disease, or Chronic Kidney Disease
Brief Title: Real-world Treatment of H. Pylori Eradication in Patients with Comorbidity
Acronym: Real-world_Hp
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: B-ER-109-072
Record Dates: First submitted 2022-07-24; First posted 2022-07-27 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2023-10

CONDITIONS: Helicobacter Pylori Infection; Comorbidities and Coexisting Conditions; Real-world Outcome; Medication Adherence; Patient Compliance; Patient Dropouts
Keywords: Helicobacter pylori; Comorbidity; Patient dropouts; Medication adherence
MeSH Terms: conditions — Medication Adherence; Patient Compliance; Patient Dropouts

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- The Charlson scores >= 2: Patients who are >= 20 years and diagnosed with H. pylori infection either by rapid urease test or by histology from January 1, 2012 to December 31, 2019 are reviewed retrospectively. Patients are excluded if they ever received H. pylori eradication before. Patient characteristics, including age, sex, and the parameters of the Charlson scores, are recorded and analyzed. Moreover, the tablet number and varieties of medications patients took for underlying diseases are also recorded. If the patients' Charlson scores >= 2, they are divided into the Charlson scores >= 2 group.
  Interventions: Drug: The sequential therapy; Drug: The triple therapy; Drug: The hybrid therapy; Drug: The concomitant therapy; Drug: Bismuth-based quadruple therapy
- The Charlson scores < 2: Patients who are >= 20 years and diagnosed with H. pylori infection either by rapid urease test or by histology from January 1, 2012 to December 31, 2019 are reviewed retrospectively. Patients are excluded if they ever received H. pylori eradication before. Patient characteristics, including age, sex, and the parameters of the Charlson scores, are recorded and analyzed. Moreover, the tablet number and varieties of medications patients took for underlying diseases are also recorded. If the patients' Charlson scores < 2, they are divided into the Charlson scores < 2 group.
  Interventions: Drug: The sequential therapy; Drug: The triple therapy; Drug: The hybrid therapy; Drug: The concomitant therapy; Drug: Bismuth-based quadruple therapy

INTERVENTIONS:
Drug: The sequential therapy — Proton pump inhibitors and amoxicillin for the first 5 or 7 days and sequent proton pump inhibitors, clarithromycin, and metronidazole for the next 5 or 7 days
Drug: The triple therapy — Proton pump inhibitors, amoxicillin, and clarithromycin for 7, 10, or 14 days.
Drug: The hybrid therapy — Proton pump inhibitors and amoxicillin starting from the 1st day and for a total of 10 or 14 days, and clarithromycin, and metronidazole starting from the 8th day and for a total of 7 days .
Drug: The concomitant therapy — Proton pump inhibitors, amoxicillin, clarithromycin, and metronidazole for a total of 7 or 14 days
Drug: Bismuth-based quadruple therapy — Proton pump inhibitors, bismuth, tetracycline, and metronidazole for a total of 10 or 14 days

SUMMARY:
Most of the studies of H. pylori eradication were conducted in academic institutes and designed to enrolled patients who did not have comorbidities. However, patients in the real world may comorbid with diabetes, chronic obstructive pulmonary disease, cirrhosis, chronic kidney diseases, or others. We hypothesize that the eradication rate of H. pylori in patients with comorbidity is poor because they may be infected with antibiotics-resistant H. pylori strains or have poor medication adherence. Here, we design a study, which focus on the H. pylori eradication rates by the various regimens in the real world, especially for those with high Charlson scores. It is presumed that our data will be helpful with regard to treating such patients with H. pylori eradication in the clinical scenario.

DETAILED DESCRIPTION:
There is a challenge for eradicating Helicobacter pylori (H. pylori) because the resistant strains of H. pylori are increasing. In order to overcome the challenge, the new regimens are developed, including 14-day triple therapy, 10-day sequential therapy, 10-day bismuth-based quadruple therapy, 10-day concomitant therapy, or 14-day hybrid therapy, which have 84%~99% of successful eradication rates. Additionally, there is a new challenge, i.e., worldwide population aging and increases in the proportion of patients with comorbidity. Most of the studies of H. pylori eradication were conducted in academic institutes and designed to enrolled patients who did not have comorbidities. However, patients in the real world may comorbid with diabetes, chronic obstructive pulmonary disease, cirrhosis, chronic kidney diseases, or others. Our previous study showed that the eradication rate of 10-day clarithromycin-based sequential therapy was 81% in diabetic patients, lower than 87% in non-diabetic patients in other study. Therefore, we hypothesize that the eradication rate of H. pylori in patients with comorbidity is poor because they may be infected with antibiotics-resistant H. pylori strains or have poor medication adherence. The former is because patients may use macrolides because of chronic obstructive pulmonary disease with airway infection, for example. The latter is because the regimen of H. pylori eradication is complex, either three or four varieties of pills and dosage intervals for administration. Moreover, the patients may have taken many other medications for their underline comorbidity. These medications may have drug-drug interaction with the H. pylori eradication regimen or make the medication adherence poor. Most of studies which were conducted in academic institutes, patients took the H. pylori eradication regimen under the study staffs' instruction and monitor; however, in the real world, their medication adherence for H. pylori eradication may be compromised. Here, we design a study, which focus on the H. pylori eradication rates by the various regimens in the real world, especially for those with high Charlson scores. It is presumed that our data will be helpful with regard to treating such patients with H. pylori eradication in the clinical scenario.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are >= 20 years and received the therapy for H. pylori eradication from January 1, 2012 to December 31, 2019 are reviewed retrospectively. The regimens include 10- or 14-day sequential therapy, 7-, 10-, or 14-day triple therapy, 10- or 14-day hybrid therapy, 7- or 14-day concomitant therapy, 10- or 14-day bismuth-based quadruple therapy.

Exclusion Criteria:

* Patients are excluded if they ever received H. pylori eradication before.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is conducted at the outpatient department of National Cheng Kung University Hospital in Tainan, Taiwan. Patients who are diagnosed with H. pylori infection and receive H. pylori eradication in the hospital are the candidates to be reviewed.
Sampling Method: Probability Sample
Enrollment: 1053 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The eradication rate by the intention-to-treat analysis | At least six weeks after the completion of H. pylori eradication
  Successful H. pylori eradication is confirmed by the 13C-urea breath test, rapid urease test, or H. pylori stool antigen test. All the reviewed patients are analyzed for intention-to-treat of H. pylori eradication.
The eradication rate by the per-protocol analysis | At least six weeks after the completion of H. pylori eradication
  Successful H. pylori eradication is confirmed by the 13C-urea breath test, rapid urease test, or H. pylori stool antigen test. Patients who do not complete the regimens or do not receive the confirmation of successful H. pylori eradication by the 13C-urea breath test, rapid urease test, or H. pylori stool antigen test are excluded from the per-protocol analysis.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan, Taiwan
  - Helicobacter pylori study group, National Cheng Kung University Hospital, Tainan

IPD SHARING:
Plan to Share IPD: No